CLINICAL TRIAL: NCT03413176
Title: Evaluation of Reporting of VEGF Inhibitors Associated Cardiovasclular Adverse reactioNs Using International Pharmacovigilance Database.
Brief Title: Evaluation of Reporting of Vascular Endothelial Growth Factor and Vascular Endothelial Growth Factor Receptor Inhibitors Associated Cardiovascular Adverse reactioN.
Acronym: VEGAN
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, MD, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-18-02
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Cardiac Complication; Vascular Diseases
Keywords: VEGFR; VEGF; antiangiogenics; angiogenesis
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Cardiac complication induced by VEGF/VEGFR inhibitor — Case reported in the World Health Organization (WHO) of cardiac complication of patient treated by AAs, with a chronology compatible with the drug toxicity

SUMMARY:
Antiangiogenics (AAs) which are vascular endothelial growth factor (VEGF) or VEGF receptor (VEGFR) inhibitors might have high grade adverse events (AEs) on the cardio-vascular system. This study investigates reports of cardio-vascular toxicity with treatment including VEGF and VEGFR inhibitors using the World Health Organization (WHO) database VigiBase.

DETAILED DESCRIPTION:
AAs have dramatically improved clinical outcomes in multiple cancer types and are increasingly being tested in earlier disease settings and used in combination. However, AEs can occur. Here the investigators use VigiBase (http://www.vigiaccess.org/), the World Health Organization (WHO) database of individual safety case reports, to identify cases of cardiovascular adverse drug reaction following treatment with AAs.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the World Health Organization (WHO) database of individual safety case reports to 01/01/2018
* Adverse event reported were including the MedDRA terms: Cardiac disorders (SOC), Vascular disorders (SOC), Sudden death (PT)
* Patients treated with antiangiogenics included in the following list:

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with an AA for a cancer
Sampling Method: Non-Probability Sample
Enrollment: 150000 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Cardio-vascular toxicity of AAs | Case reported in the World Health Organization (WHO) database of individual safety case reports to 01/01/2018
  Identification and report of the cardio-vascular toxicity of AAs. The research includes the report with MedDRA terms: SOC Cardiac Disorders, SOC Vascular Disorders, Sudden death (PT). Drugs investigated are: sorafenib, sunitinib, pazopanib, vandetanib, axitinib, regorafenib, nintedanib, lenvatinib, ceritinib, bevacizumab, ramucirumab, aflibercept.

SECONDARY OUTCOMES:
Causality assessment of reported cardiovascular events according to the WHO system | Case reported in the World Health Organization (WHO) database of individual safety case reports to 01/01/2018
Description of the type of cardiotoxicity depending on the category of AAs | Case reported in the World Health Organization (WHO) database of individual safety case reports to 01/01/2018
Description of the duration of treatment when the toxicity happens (role of cumulative dose) | Case reported in the World Health Organization (WHO) database of individual safety case reports to 01/01/2018
Description of the drug-drug interactions associated with adverse events | Case reported in the World Health Organization (WHO) database of individual safety case reports to 01/01/2018
Description of the pathologies (cancer) for which the incriminated drugs have been prescribed | Case reported in the World Health Organization (WHO) database of individual safety case reports to 01/01/2018
Description of the population of patients having a cardio-vascular adverse event | Case reported in the World Health Organization (WHO) database of individual safety case reports to 01/01/2018

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM., Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alexandre J, Moslehi JJ, Bersell KR, Funck-Brentano C, Roden DM, Salem JE. Anticancer drug-induced cardiac rhythm disorders: Current knowledge and basic underlying mechanisms. Pharmacol Ther. 2018 Sep;189:89-103. doi: 10.1016/j.pharmthera.2018.04.009. Epub 2018 Apr 24. PMID 29698683
- [Background] Gougis P, Wassermann J, Spano JP, Keynan N, Funck-Brentano C, Salem JE. Clinical pharmacology of anti-angiogenic drugs in oncology. Crit Rev Oncol Hematol. 2017 Nov;119:75-93. doi: 10.1016/j.critrevonc.2017.08.010. Epub 2017 Sep 1. PMID 28916378